CLINICAL TRIAL: NCT00553514
Title: A Phase II, Multicentre, Randomised, Assessor-blinded, Active-comparator, Parallel-group Dose Finding Trial to Evaluate AS900672-enriched Versus Follitropin Alfa (GONAL-f®) in Oligo-anovulatory Infertile Women Undergoing Ovulation Induction (OI)
Brief Title: AS900672-Enriched in Ovulation Induction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated after Merck Serono had taken the decision not to pursue the development of AS900672-enriched in ovulation induction
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27818
Record Dates: First submitted 2007-11-01; First posted 2007-11-05 (Estimated); Results first posted 2013-07-25 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Ovulation Induction
Keywords: Infertility; Oligo-anovulation; GONAL-f®; AS900672-Enriched; hyperglycosylated recombinant human follicle stimulating hormone (r-hFSH)
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; Follicle Stimulating Hormone; Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (5):
- AS900672-Enriched 10 mcg (Experimental)
  Interventions: Drug: AS900672-Enriched 10 microgram (mcg); Drug: Follitropin alfa 75 international unit (IU); Drug: Recombinant human chorionic gonadotropin (r-hCG)
- AS900672-Enriched 20 mcg (Experimental)
  Interventions: Drug: AS900672-Enriched 20 mcg; Drug: Follitropin alfa 75 international unit (IU); Drug: Recombinant human chorionic gonadotropin (r-hCG)
- AS900672-Enriched 30 mcg (Experimental)
  Interventions: Drug: AS900672-Enriched 30 mcg; Drug: Follitropin alfa 75 international unit (IU); Drug: Recombinant human chorionic gonadotropin (r-hCG)
- AS900672-Enriched 40 mcg (Experimental)
  Interventions: Drug: AS900672-Enriched 40 mcg; Drug: Follitropin alfa 75 international unit (IU); Drug: Recombinant human chorionic gonadotropin (r-hCG)
- Follitropin alfa 75 IU (Active Comparator)
  Interventions: Drug: Follitropin alfa 75 international unit (IU); Drug: Recombinant human chorionic gonadotropin (r-hCG)

INTERVENTIONS:
Drug: AS900672-Enriched 10 microgram (mcg) — Single injection of AS900672-Enriched (hyperglycosylated recombinant human follicle stimulating hormone [r-hFSH]), 10 mcg will be administered subcutaneously on Stimulation Day 1 (S1). Duration of treatment cycle will be up to adequate follicular response received or maximum of 14 days.
  Other Names: Hyperglycosylated r-hFSH
  Arms: AS900672-Enriched 10 mcg
Drug: AS900672-Enriched 20 mcg — Single injection of AS900672-Enriched (hyperglycosylated r-hFSH), 20 mcg will be administered subcutaneously on S1. Duration of treatment cycle will be up to adequate follicular response received or maximum of 14 days.
  Other Names: Hyperglycosylated r-hFSH
  Arms: AS900672-Enriched 20 mcg
Drug: AS900672-Enriched 30 mcg — Single injection of AS900672-Enriched (hyperglycosylated r-hFSH), 30 mcg will be administered subcutaneously on S1. Duration of treatment cycle will be up to adequate follicular response received or maximum of 14 days.
  Other Names: Hyperglycosylated r-hFSH
  Arms: AS900672-Enriched 30 mcg
Drug: AS900672-Enriched 40 mcg — Single injection of AS900672-Enriched (hyperglycosylated r-hFSH), 40 mcg will be administered subcutaneously on S1. Duration of treatment cycle will be up to adequate follicular response received or maximum of 14 days.
  Other Names: Hyperglycosylated r-hFSH
  Arms: AS900672-Enriched 40 mcg
Drug: Follitropin alfa 75 international unit (IU) — Follitropin alfa (Gonal-f®) 75 IU will be administered subcutaneously once daily from S1 up to Stimulation Day 14 (S14) based upon ovarian response, until recombinant human chorionic gonadotropin (r-hCG) administration day. Subjects who will be receiving AS900672-Enriched 10, 20, 30 and 40 mcg will also receive daily dose of follitropin alfa 75 IU subcutaneously from Stimulation Day 7 (S7) up to S14. Duration of treatment cycle will be up to adequate follicular response received or maximum of 14 days.
  Other Names: Gonal-f®; Follicle stimulating hormone (FSH)
Drug: Recombinant human chorionic gonadotropin (r-hCG) — Recombinant human chorionic gonadotropin (r-hCG) will be administered as a single dose of 250 mcg subcutaneously, when follicular response is adequate (that is, less than or equal to [=<] 3 follicles with a mean diameter of greater than or equal to [>=] 14 millimeter [mm], and one or two of these follicles with a diameter of >= 17 mm).

SUMMARY:
This is a Phase 2, interventional, multi-center, randomized, assessor-blind, active-comparator, dose-finding study to evaluate a new investigational long-acting follicle stimulating hormone (FSH) in oligo-anovulatory women undergoing ovulation induction (OI). This study will compare 4 doses of the investigational drug versus a currently marketed drug follitropin alfa (Gonal-f ®) prefilled pen with regards to ovulation rate.

DETAILED DESCRIPTION:
The study was terminated after Merck Serono had taken the decision not to pursue the development of AS900672-enriched in ovulation induction (OI). This decision was not related to any safety or efficacy concerns over the use of AS900672-Enriched in OI.

ELIGIBILITY:
Inclusion Criteria:

* Oligo-anovulation defined by a menstrual period of 35 days to 6 months
* Spontaneous menses or a positive response to progestin within the prior 6 months or response to clomiphene citrate evidenced by ovulation within the prior 6 months
* Age between 18 and 36 years, inclusive, at time of informed consent signature
* Body mass index (BMI) 18 to 30 kilogram per square meter (kg/m^2), inclusive
* No clinically significant abnormalities in serum thyroid stimulating hormone (TSH), dehydroepiandrosterone (DHEA-S), prolactin, and FSH levels in the early follicular phase. Subjects low TSH level who receive replacement therapy could be enrolled at the discretion of the investigator if local laboratory results (thyroxine [T4]) demonstrated satisfactory thyroid function. Subjects receiving stable dose of dopamine agonists could be enrolled at the discretion of the investigator if local laboratory results demonstrated adequate control of prolactin levels
* No clinically significant abnormalities in fasting glucose and fasting insulin levels
* Normal uterine cavity and presence of at least one ovary with ipsilateral patent fallopian tube, as determined by means of hysterosalpingography, laparoscopy, hysteroscopy or combination of these procedures within the prior 3 years
* Papanicolaou (PAP) smear test without clinically significant abnormalities within 6 months prior to the first screening procedure. If PAP smear is not done, it must be performed as part of screening procedures
* Negative pregnancy test prior to randomization
* Male partner with semen analysis demonstrating adequacy for insemination via intercourse and/or intrauterine insemination (IUI) within 6 months prior to the first screening procedure. If semen analysis is not done, it must be performed as part of screening procedures
* Willing and able to comply with all protocol procedures, including pregnancy and neonatal follow-up
* Voluntary provision of written informed consent, prior to any trial-related procedure that is not part of normal medical care, with the understanding that the subject could withdraw consent at any time without prejudice to her future medical care, including willingness to provide follow-up information on babies born as part of this trial

Exclusion Criteria:

* History of >=2 consecutive gonadotrophin stimulation cycles that did not lead to ovulation
* History of clomiphene citrate stimulation cycles of which none lead to ovulation
* Prior excessive response to gonadotrophin stimulation, defined as the development of at least 4 mature follicles (greater than [>]17 mm) or cancellation of the OI cycle due to excessive follicular response after treatment with FSH at a dose of less than 75 IU/day
* Previous severe ovarian hyperstimulation syndrome (OHSS)
* Administration of any gonadotrophin, clomiphene citrate, gonadotrophin releasing hormone (GnRH) analogue, tamoxifen or aromatase inhibitors within the prior 30 days
* Laparoscopic ovarian drilling and/or ovarian cauterization within the prior 6 months
* Any contraindication to pregnancy and/or to carrying pregnancy to term
* A clinical pregnancy that ended in a miscarriage within the prior 3 months
* History of >=3 consecutive miscarriages, due to any cause
* Abnormal gynecological bleeding of undetermined origin
* Clinically significant abnormal findings of the uterine cavity evident on a transvaginal pelvic ultrasound performed during screening
* Presence of endometriosis, Grade III - IV or requiring treatment
* Ovarian cyst with a mean diameter of >25 mm on the day of randomization
* History or suspicion of ovarian, uterine or mammary cancer
* Adrenal congenital hyperplasia, partial or complete enzymatic block
* Use of metformin or other insulin sensitizing agents related to infertility within the prior 2 months
* Known allergy or hypersensitivity to human gonadotrophin preparations or to compounds that are structurally similar to any of the other medications administered during the trial
* Any contra-indication to gonadotrophin therapy
* Known or suspected infection with human immunodeficiency virus (HIV), Hepatitis B or C in the trial subject or her male partner
* Any active substance abuse or history of drug, medication or alcohol abuse within 5 years
* Smoker consuming more than 5 cigarettes per day
* Serum testosterone (central laboratory) that is suggestive of ovarian tumor
* Previously randomized in this trial or participation in another investigational drug clinical trial within the prior 3 months
* Any medical condition, which in the judgment of the investigator may interfere with the absorption, distribution, metabolism or excretion of r-hFSH
* Clinically significant concurrent disease (including diabetes mellitus and autoimmune diseases) that would compromise subject safety or interfere with the study assessments or clinically significant abnormal laboratory finding

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pellicer, Professor Dr, Principal Investigator — IVI Valencia
Locations (1):
- Merck Serono S.A., Geneva, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- AS900672-Enriched 10 Mcg: Single injection of AS900672-Enriched (hyperglycosylated recombinant human follicle stimulating hormone [r-hFSH]), 10 microgram (mcg) administered subcutaneously on Stimulation day 1 (S1) followed by a daily dose of follitropin alfa 75 international unit (IU) subcutaneously starting from Stimulation Day 7 (S7) up to Stimulation Day 14 (S14) based upon ovarian response, until recombinant human chorionic gonadotropin (r-hCG) administration day. When follicular response was adequate (that is, less than or equal to [=<] 3 follicles with a mean diameter of greater than or equal to [>=] 14 millimeter [mm], and one or two of these follicles with a diameter of >= 17 mm), ovulation was triggered by single 250 mcg subcutaneous r-hCG injection. Duration of treatment cycle was up to adequate follicular response received or maximum of 14 days.
- AS900672-Enriched 20 Mcg: Single injection of AS900672-Enriched (hyperglycosylated r-hFSH), 20 mcg administered subcutaneously on S1 followed by a daily dose of follitropin alfa 75 IU subcutaneously starting from S7 up to S14 based upon ovarian response, until r-hCG administration day. When follicular response was adequate (that is, =< 3 follicles with a mean diameter of >=14 mm, and one or two of these follicles with a diameter of >=17 mm), ovulation was triggered by single 250 mcg subcutaneous r-hCG injection. Duration of treatment cycle was up to adequate follicular response received or maximum of 14 days.
- AS900672-Enriched 30 Mcg: Single injection of AS900672-Enriched (hyperglycosylated r-hFSH), 30 mcg administered subcutaneously on S1 followed by a daily dose of follitropin alfa 75 IU subcutaneously starting from S7 up to S14 based upon ovarian response, until r-hCG administration day. When follicular response was adequate (that is, =< 3 follicles with a mean diameter of >=14 mm, and one or two of these follicles with a diameter of >=17 mm), ovulation was triggered by single 250 mcg subcutaneous r-hCG injection. Duration of treatment cycle was up to adequate follicular response received or maximum of 14 days.
- AS900672-Enriched 40 Mcg: Single injection of AS900672-Enriched (hyperglycosylated r-hFSH), 40 mcg administered subcutaneously on S1 followed by a daily dose of follitropin alfa 75 IU subcutaneously starting from S7 up to S14 based upon ovarian response, until r-hCG administration day. When follicular response was adequate (that is, =< 3 follicles with a mean diameter of >=14 mm, and one or two of these follicles with a diameter of >=17 mm), ovulation was triggered by single 250 mcg subcutaneous r-hCG injection. Duration of treatment cycle was up to adequate follicular response received or maximum of 14 days.
- Follitropin Alfa 75 IU: Follitropin alfa (Gonal-f®) 75 IU administered subcutaneously once daily from S1 up to S14 based upon ovarian response, until r-hCG administration day. When follicular response was adequate (that is, =< 3 follicles with a mean diameter of >=14 mm, and one or two of these follicles with a diameter of >=17 mm), ovulation was triggered by single 250 mcg subcutaneous r-hCG injection. Duration of treatment cycle was up to adequate follicular response received or maximum of 14 days.
Period: Overall Study
Arm/Group | AS900672-Enriched 10 Mcg | AS900672-Enriched 20 Mcg | AS900672-Enriched 30 Mcg | AS900672-Enriched 40 Mcg | Follitropin Alfa 75 IU
Started | 14 | 14 | 15 | 13 | 15
Completed | 6 | 6 | 9 | 6 | 8
Not Completed | 8 | 8 | 6 | 7 | 7
Not completed — Protocol deviation | 0 | 0 | 0 | 1 | 0
Not completed — Lack of ovarian response | 4 | 5 | 5 | 5 | 6
Not completed — Ovarian hyperstimulation syndrome risk | 3 | 0 | 1 | 0 | 0
Not completed — Risk of multiple pregnancy | 0 | 2 | 0 | 1 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AS900672-Enriched 10 Mcg | AS900672-Enriched 20 Mcg | AS900672-Enriched 30 Mcg | AS900672-Enriched 40 Mcg | Follitropin Alfa 75 IU | Total
Number analyzed (Participants) | 14 | 14 | 15 | 13 | 15 | 71
Age, Continuous [Median (Full Range); unit: years] | 29.5 [23 to 36] | 31.5 [23 to 36] | 28.0 [26 to 35] | 30.0 [23 to 36] | 30.0 [23 to 34] | 30 [23 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 15 | 13 | 15 | 71
  Male | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Ovulation
Description: Ovulation was defined as a mid-luteal phase progesterone (P4) level >= 30 nanomole per liter (nmol/L) (10 nanogram per milliliter [ng/mL]). In the absence of a positive progesterone response, clinical pregnancy was also considered as evidence of ovulation.
Time Frame: Mid-luteal phase progesterone assessed 5-10 days or clinical pregnancy 35-42 days after recombinant human chorionic gonadotropin (r-hCG) administration day (end of stimulation cycle [approximately 14 days])
Population: Per Protocol (PP) population included all the randomized participants who were without a medically relevant protocol deviation. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | AS900672-Enriched 10 Mcg | AS900672-Enriched 20 Mcg | AS900672-Enriched 30 Mcg | AS900672-Enriched 40 Mcg | Follitropin Alfa 75 IU
Number analyzed (Participants) | 13 | 13 | 13 | 12 | 13
Percentage of participants | 46.2 | 46.2 | 38.5 | 33.3 | 53.8

2. Secondary Outcome: Percentage of Participants With Clinical Pregnancy
Description: Clinical pregnancy was defined as the presence of one or more fetal sacs with fetal heart activity on the Day 35-42 post r-hCG ultrasound examination.
Time Frame: Day 35-42 post r-hCG administration day (end of stimulation cycle [approximately 14 days])
Population: PP population included all the randomized participants who were without a medically relevant protocol deviation. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | AS900672-Enriched 10 Mcg | AS900672-Enriched 20 Mcg | AS900672-Enriched 30 Mcg | AS900672-Enriched 40 Mcg | Follitropin Alfa 75 IU
Number analyzed (Participants) | 13 | 13 | 13 | 12 | 13
Percentage of participants | 23.1 | 0.0 | 7.7 | 16.7 | 0.0

3. Secondary Outcome: Duration of Ovarian Stimulation
Description: Ovarian stimulation included from first dose of study drug on S1 until day on which r-hCG was administered (r-hCG day).
Time Frame: Stimulation Day 1 (S1) up to r-hCG administration day (end of stimulation cycle [approximately 14 days])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AS900672-Enriched 10 Mcg | AS900672-Enriched 20 Mcg | AS900672-Enriched 30 Mcg | AS900672-Enriched 40 Mcg | Follitropin Alfa 75 IU
Number analyzed (Participants) | 13 | 13 | 13 | 12 | 13
Days | 10.0 (5.3) | 11.8 (3.4) | 14.0 (1.4) | 10.8 (3.7) | 10.6 (3.2)

4. Secondary Outcome: Duration of Supplemental Follitropin Alfa Treatment
Time Frame: Stimulation Day 7 (S7) up to r-hCG administration day (end of stimulation cycle [approximately 14 days])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AS900672-Enriched 10 Mcg | AS900672-Enriched 20 Mcg | AS900672-Enriched 30 Mcg | AS900672-Enriched 40 Mcg | Follitropin Alfa 75 IU
Number analyzed (Participants) | 10 | 12 | 13 | 11 | 11
Days | 6.6 (1.4) | 6.6 (1.4) | 7.7 (1.5) | 5.6 (2.2) | 5.5 (2.7)

5. Secondary Outcome: Cumulative Dose of Supplemental Follitropin Alfa Administered
Time Frame: Stimulation Day 7 (S7) up to r-hCG administration day (end of stimulation cycle [approximately 14 days])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | AS900672-Enriched 10 Mcg | AS900672-Enriched 20 Mcg | AS900672-Enriched 30 Mcg | AS900672-Enriched 40 Mcg | Follitropin Alfa 75 IU
Number analyzed (Participants) | 10 | 12 | 13 | 11 | 10
IU | 476.3 (122.5) | 493.8 (108.3) | 556.7 (134.2) | 398.9 (167.9) | 397.5 (226.5)

6. Secondary Outcome: Number of Follicles With Mean Diameter Less Than (<) 11 Millimeter (mm) and Greater Than or Equal to (>=) 11 mm
Time Frame: Stimulation Day 5 (S5), S7 and r-hCG administration day (end of stimulation cycle [approximately 14 days])
Population: PP population included all the randomized participants who were without a medically relevant protocol deviation. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure. 'n' signifies number of participants who were evaluable for specified categories at different time points.
Measure: Mean (Standard Deviation); unit: Follicles
Arm/Group | AS900672-Enriched 10 Mcg | AS900672-Enriched 20 Mcg | AS900672-Enriched 30 Mcg | AS900672-Enriched 40 Mcg | Follitropin Alfa 75 IU
Number analyzed (Participants) | 12 | 12 | 13 | 12 | 13
Follicles
  < 11 mm on S5 (n=12,12,12,12,13) | 23.6 (13.8) | 28.7 (29.4) | 23.2 (6.7) | 20.9 (16.7) | 21.3 (13.7)
  < 11 mm on S7 (n=12,12,13,12,12) | 22.8 (12.6) | 27.2 (30.9) | 21.0 (8.9) | 21.3 (17.3) | 22.0 (16.7)
  < 11 mm on r-hCG Day (n=5,6,7,6,7) | 15.6 (7.3) | 11.7 (9.2) | 18.4 (12.1) | 18.7 (15.0) | 14.9 (12.4)
  >= 11 mm on S5 (n=12,8,7,11,8) | 1.5 (2.2) | 0.0 (0.0) | 1.6 (1.9) | 2.8 (3.1) | 0.8 (0.9)
  >= 11 mm on S7 (n=11,9,7,11,11) | 3.4 (6.2) | 0.2 (0.7) | 2.6 (3.5) | 2.8 (2.4) | 1.8 (2.3)
  >= 11 mm on r-hCG Day (n=5,6,8,6,8) | 2.6 (0.9) | 2.5 (1.9) | 2.5 (1.3) | 1.8 (0.8) | 2.9 (1.8)

ADVERSE EVENTS:
Time Frame: Stimulation Day 1 (S1) up to Day 35-42 post r-hCG administration day (end of stimulation cycle [approximately 14 days])
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an investigational medicinal product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | AS900672-Enriched 10 Mcg | AS900672-Enriched 20 Mcg | AS900672-Enriched 30 Mcg | AS900672-Enriched 40 Mcg | Follitropin Alfa 75 IU
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/15 | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 7/14 | 3/14 | 6/15 | 4/13 | 7/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AS900672-Enriched 10 Mcg (N=14) | AS900672-Enriched 20 Mcg (N=14) | AS900672-Enriched 30 Mcg (N=15) | AS900672-Enriched 40 Mcg (N=13) | Follitropin Alfa 75 IU (N=15)
Headache (Nervous system disorders) | 2 | 1 | 3 | 3 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Adnexa uteri pain (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated after Merck Serono had taken the decision not to pursue the development of AS900672-enriched in ovulation induction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other